CLINICAL TRIAL: NCT04029454
Title: Neovac 2 Burkina Faso: Impact of the Integration of Hepatitis B Birth Dose Vaccine Into the Infant Immunization Schedule: a Mixed Methods Study Including a Cluster-randomized Trial, an Anthropological Study and an Economic Evaluation
Brief Title: Neovac 2 Burkina Faso: Impact of the Integration of Hepatitis B Birth Dose Vaccine Into the Infant Immunization Schedule
Acronym: NEOVAC2BK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Pasteur (Industry)
Collaborators: Agence de Médecine Préventive, France (Other); Centre Muraz (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Gilead Sciences (Industry); Abbott (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 2017-083
Record Dates: First submitted 2019-06-05; First posted 2019-07-23 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Hepatitis B
Keywords: Infectious Disease Transmission, Vertical; immunization programs
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Intervention Model Description: Pragmatic Stepped-wedge cluster randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention period (Experimental): Intervention : birth dose vaccination against hepatitis B strategy Birth dose of vaccine against hepatitis B + routine Expended Programme on Imunisation (EPI) vaccination schedule starting at 8 weeks of life
  Interventions: Biological: birth dose vaccination against hepatitis B strategy
- Control period (No Intervention): Routine Expended Programme on Imunisation (EPI) vaccination schedule starting at 8 weeks of life

INTERVENTIONS:
Biological: birth dose vaccination against hepatitis B strategy — Complex intervention targeting healthcare workers and involving:
  * training on hepatitis B awareness and management
  * training on EPI vaccination and cold chain
  * training on the modalities for the birth dose administration
  * the use of a monovalent unidose vaccine against Hepatitis B
  Arms: Intervention period

SUMMARY:
Hepatitis B virus (HBV) infection is an important global health problem, and the WHO adopted a strategy to eliminate HBV infection as a public health threat by the year 2030. In order to eliminate, it is critical to prevent the mother-to-child transmission (MTCT) of hepatitis B. Since 2009, the WHO recommends to administer hepatitis B vaccine within 24 hours of birth to prevent MTCT.2 However, in Africa, the majority of countries provide hepatitis B vaccine as a combined vaccine (pentavalent or hexavalent) at the age of 6-10-14 weeks or 8-12-16 weeks after the birth, and only 10 sub-Saharan African countries integrated birth dose vaccine into their national immunization program. This is because, the GAVI, the Vaccine Alliance, does not support monovalent hepatitis B vaccine, and also about half of babies in Africa are born at home without the immediate access to vaccination. Moreover, the evidence base to support this WHO's recommendation to start immunizing immediately at birth, rather than later at 6-8 weeks of life, is not strong.

Through a multidisciplinary approach comprising epidemiological, anthropological and economic components, the primary objective of the study is to measure the impact of the introduction of birth dose hepatitis B vaccine into the infant immunization program in Burkina Faso.

Expected results will be to develop strong evidence base (effectiveness & cost-effectiveness) to recommend the integration of birth dose hepatitis B vaccine into the current vaccination schedule (8-12-16 weeks as a combined vaccine), to facilitate the Burkinabé Government to include the birth dose hepatitis B vaccine in their national vaccination program, to inform other African countries which have not yet integrated the birth dose hepatitis B vaccine in their national program and to imply whether additional strategy (e.g., maternal screening and antiviral therapy during pregnancy) might be necessary in order to eliminate the risk of mother-to-child transmission of hepatitis B.

DETAILED DESCRIPTION:
The study combines mixed methods to achieve its aim of evaluating the impact of the introduction of birth dose hepatitis B vaccine into the infant immunisation program in Burkina Faso. It is composed of 4 components:

Workpackage (WP1): Stepped Wedge Cluster randomized controlled trial:

* to measure the impact of the introduction of birth dose hepatitis B vaccine into the infant immunization program on the mother-to-child transmission (primary objective)
* To examine a dose-dependent effect of hepatitis B vaccine (according to the total number of doses from one to four doses)
* To examine a time-dependent effect of the first dose of hepatitis B vaccine
* To study the impact of birth dose vaccine in infants aged at 9 months according to maternal HBsAg and HBeAg status
* To compare immunological responses in both groups by titration of anti-HBs antibodies in children at 9 months
* To describe vaccine coverage and its timeliness of birth dose hepatitis B vaccine and other routine infant vaccines in Burkina Faso
* To estimate the prevalence of HBV infection in mothers of 9-month-old children

WP2: Anthropological study • To evaluate the acceptability of healthcare workers and people in the community about the integration of hepatitis B birth dose vaccine in the infant vaccination program in Burkina Faso

WP3: Economic evaluation

* To evaluate the cost-effectiveness of the integration of hepatitis B birth dose vaccine in the infant vaccination program, compared to the conventional vaccine schedule (8-12-16 weeks) in Burkina Faso
* To evaluate the diagnostic performance of low-cost HBV markers to identify women at high risk of mother-to-child transmission in low-income countries

WP4: Virological evaluation

• To evaluate the diagnostic performance of low-cost HBV markers to identify women at high risk of mother-to-child transmission in low-income countries

All the pregnant women attending the antenatal care in the rural health centres of two health districts (Dafra and Dô) in Hauts Bassins Region in Burkina Faso, and their infants will be asked to participate.

Practical sequence of the cluster randomised trial. Even though the evidence is weak and the implementation has been suboptimal, the WHO currently recommends the universal administration of hepatitis B vaccine at birth. For this reason, a "stepped-wedge" design rather than a parallel group design has been selected. Of 24 rural health centers (Centre de santé et de promotion sociale : CSPS) in the districts of Dafra and Dô, introduce monovalent birth dose vaccine will be introduced in a phased manner on a centre by centre basis until all the 24 CSPSs integrate the birth dose vaccines in the program. The rural area of these districts were selected given the proximity to our collaborative study center (Centre Muraz and AMP in Bobo Dioulasso). One of the 24 centers will be randomly selected as the first one to start integrating the birth dose in the program. Then, four weeks later, the second center will be randomly selected to start providing the birth dose vaccine. This will be continued until all 24 CSPSs integrate birth dose vaccine in the program. At the end, this study design will generate two groups of infants in the study area during the study period: those born in centres which already implemented birth dose vaccine, and those born before the introduction of this vaccine.

Informed consent will be obtained from pregnant women who visited routine antenatal care. Subsequently, babies born in a CSPS which is in the intervention period will receive birth dose vaccine whilst those born in a CSPS which is in the control period will not receive the birth dose. For those born at home in the intervention period will receive the monovalent hepatitis B vaccine at the first contact with CSPS, until 8 weeks after the birth when the first dose of pentavalent vaccine (DPT-Hib-HepB) is scheduled. All the infants, irrespective of study period, will receive three doses of pentavalent vaccine as scheduled in the national immunization program.

Case report forms will be used (CRFs to collect basic demographic data of mothers and infants; time and place of birth; type of vaccines administered and its date Laboratory data: HBsAg for all infants and mothers; HBV DNA, HBeAg, AST/ALT for infants and mothers tested positive for HBsAg; anti-HBs for infants tested negative for HBsAg Paper CRFs filled by healthcare workers will be transferred to the study centre (AMP/Centre Muraz). The data will be entered independently by two operators to electronic database (RedCAP) that will be developed on the secured server of the Institut Pasteur.

The risk of HBV infection (HBsAg-positivity) in infants at the age of 9 months between two groups will be compared using an intention-to-treat analysis, in order to assess the effectiveness of adding birth dose vaccine compared to the current vaccine schedule in preventing the mother-to-child transmission in Burkina Faso. To adjust for the calendar time and clustering in the data, A logistic regression model will fit with random effect for cluster and fixed effect for each step.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman
* Living in the study area
* Visited study health centre for the antenatal care or child delivery
* Provided a written informed consent

Exclusion Criteria:

* Miscarriage, abortion, stillborn, neonatal defect incompatible with life
* Any mother or child condition incompatible with the research activities

Ages: 15 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 10000 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Proportion of positive HBV infection in 9-month-old children vaccinated at birth compared to children receiving their first vaccination at 8 weeks. | at 9 months old
  Capillary blood obtained by finger-prick will be used for a rapid diagnostic test for HBsAg detection in order to identify positive hepatitis B surface antigen (HBsAg) in infants and their mother then compare immunological responses by study arm (children who received the birth dose versus those who did not receive it) on titration of anti-HBs antibodies.

SECONDARY OUTCOMES:
Prevalence rate of HBV infection in pregnancy from HBsAg and HBeAg profiles in mothers of 9-month-old children | at 9 months
  Positive hepatitis B surface antigen (capillary blood obtained by finger-prick) and positive hepatitis B e surface antigen (blood sample).
Sensibility and specificity of low-cost alternative HBV markers | 9 months after delivery
  qHBsAg, qHBeAg, RDT HBeAg, HBcrAg, and HBV LAMP results obtained with sera samples of HBsAg positive women will be compared to qPCR results as reference. Their performance (sensibility and specificity) to identify women at high risk of mother-to-child transmission (≥200 000 IU/mL) will then be calculated

CONTACTS AND LOCATIONS:
Locations (2):
- Burkina Faso (2):
  - District sanitaire de Dafra, Bobo-Dioulasso, Dafra
  - District sanitaire de Do, Bobo-Dioulasso, Do

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schweitzer A, Horn J, Mikolajczyk RT, Krause G, Ott JJ. Estimations of worldwide prevalence of chronic hepatitis B virus infection: a systematic review of data published between 1965 and 2013. Lancet. 2015 Oct 17;386(10003):1546-55. doi: 10.1016/S0140-6736(15)61412-X. Epub 2015 Jul 28. PMID 26231459
- [Background] MacLachlan JH, Cowie BC. Hepatitis B virus epidemiology. Cold Spring Harb Perspect Med. 2015 May 1;5(5):a021410. doi: 10.1101/cshperspect.a021410. PMID 25934461
- [Background] World Health Organization. Hepatitis B vaccines: WHO position paper, July 2017 - Recommendations. Vaccine. 2019 Jan 7;37(2):223-225. doi: 10.1016/j.vaccine.2017.07.046. Epub 2017 Jul 22. PMID 28743487
- [Background] Burk RD, Hwang LY, Ho GY, Shafritz DA, Beasley RP. Outcome of perinatal hepatitis B virus exposure is dependent on maternal virus load. J Infect Dis. 1994 Dec;170(6):1418-23. doi: 10.1093/infdis/170.6.1418. PMID 7995980
- [Background] Tamandjou CR, Maponga TG, Chotun N, Preiser W, Andersson MI. Is hepatitis B birth dose vaccine needed in Africa? Pan Afr Med J. 2017 Jun 22;27(Suppl 3):18. doi: 10.11604/pamj.supp.2017.27.3.11546. eCollection 2017. PMID 29296153
- [Background] Pan CQ, Zou HB, Chen Y, Zhang X, Zhang H, Li J, Duan Z. Cesarean section reduces perinatal transmission of hepatitis B virus infection from hepatitis B surface antigen-positive women to their infants. Clin Gastroenterol Hepatol. 2013 Oct;11(10):1349-55. doi: 10.1016/j.cgh.2013.04.026. Epub 2013 Apr 29. PMID 23639606
- [Background] Edmunds WJ, Medley GF, Nokes DJ, O'Callaghan CJ, Whittle HC, Hall AJ. Epidemiological patterns of hepatitis B virus (HBV) in highly endemic areas. Epidemiol Infect. 1996 Oct;117(2):313-25. doi: 10.1017/s0950268800001497. PMID 8870629
- [Background] Barin F, Perrin J, Chotard J, Denis F, N'Doye R, Diop Mar I, Chiron JP, Coursaget P, Goudeau A, Maupas P. Cross-sectional and longitudinal epidemiology of hepatitis B in Senegal. Prog Med Virol. 1981;27:148-62. No abstract available. PMID 6972051
- [Background] Kiire CF. The epidemiology and prophylaxis of hepatitis B in sub-Saharan Africa: a view from tropical and subtropical Africa. Gut. 1996;38 Suppl 2(Suppl 2):S5-12. doi: 10.1136/gut.38.suppl_2.s5. PMID 8786055
- [Background] Edmunds WJ, Medley GF, Nokes DJ, Hall AJ, Whittle HC. The influence of age on the development of the hepatitis B carrier state. Proc Biol Sci. 1993 Aug 23;253(1337):197-201. doi: 10.1098/rspb.1993.0102. PMID 8397416
- [Background] Shimakawa Y, Yan HJ, Tsuchiya N, Bottomley C, Hall AJ. Association of early age at establishment of chronic hepatitis B infection with persistent viral replication, liver cirrhosis and hepatocellular carcinoma: a systematic review. PLoS One. 2013 Jul 19;8(7):e69430. doi: 10.1371/journal.pone.0069430. Print 2013. PMID 23894479
- [Background] Shimakawa Y, Lemoine M, Bottomley C, Njai HF, Ndow G, Jatta A, Tamba S, Bojang L, Taal M, Nyan O, D'Alessandro U, Njie R, Thursz M, Hall AJ. Birth order and risk of hepatocellular carcinoma in chronic carriers of hepatitis B virus: a case-control study in The Gambia. Liver Int. 2015 Oct;35(10):2318-26. doi: 10.1111/liv.12814. Epub 2015 Mar 11. PMID 25728498
- [Background] Shimakawa Y, Lemoine M, Njai HF, Bottomley C, Ndow G, Goldin RD, Jatta A, Jeng-Barry A, Wegmuller R, Moore SE, Baldeh I, Taal M, D'Alessandro U, Whittle H, Njie R, Thursz M, Mendy M. Natural history of chronic HBV infection in West Africa: a longitudinal population-based study from The Gambia. Gut. 2016 Dec;65(12):2007-2016. doi: 10.1136/gutjnl-2015-309892. Epub 2015 Jul 16. PMID 26185161
- [Background] Feldstein LR, Mariat S, Gacic-Dobo M, Diallo MS, Conklin LM, Wallace AS. Global Routine Vaccination Coverage, 2016. MMWR Morb Mortal Wkly Rep. 2017 Nov 17;66(45):1252-1255. doi: 10.15585/mmwr.mm6645a3. PMID 29145357
- [Background] Kramvis A, Clements CJ. Implementing a birth dose of hepatitis B vaccine for home deliveries in Africa--too soon? Vaccine. 2010 Sep 7;28(39):6408-10. doi: 10.1016/j.vaccine.2010.07.042. Epub 2010 Jul 29. PMID 20673825
- [Background] Lee C, Gong Y, Brok J, Boxall EH, Gluud C. Hepatitis B immunisation for newborn infants of hepatitis B surface antigen-positive mothers. Cochrane Database Syst Rev. 2006 Apr 19;(2):CD004790. doi: 10.1002/14651858.CD004790.pub2. PMID 16625613
- [Background] Ekra D, Herbinger KH, Konate S, Leblond A, Fretz C, Cilote V, Douai C, Da Silva A, Gessner BD, Chauvin P. A non-randomized vaccine effectiveness trial of accelerated infant hepatitis B immunization schedules with a first dose at birth or age 6 weeks in Cote d'Ivoire. Vaccine. 2008 May 23;26(22):2753-61. doi: 10.1016/j.vaccine.2008.03.018. Epub 2008 Mar 31. PMID 18436354
- [Background] Marion SA, Tomm Pastore M, Pi DW, Mathias RG. Long-term follow-up of hepatitis B vaccine in infants of carrier mothers. Am J Epidemiol. 1994 Oct 15;140(8):734-46. doi: 10.1093/oxfordjournals.aje.a117321. PMID 7942775
- [Background] Pan CQ, Duan Z, Dai E, Zhang S, Han G, Wang Y, Zhang H, Zou H, Zhu B, Zhao W, Jiang H; China Study Group for the Mother-to-Child Transmission of Hepatitis B. Tenofovir to Prevent Hepatitis B Transmission in Mothers with High Viral Load. N Engl J Med. 2016 Jun 16;374(24):2324-34. doi: 10.1056/NEJMoa1508660. PMID 27305192
- [Background] Hemming K, Haines TP, Chilton PJ, Girling AJ, Lilford RJ. The stepped wedge cluster randomised trial: rationale, design, analysis, and reporting. BMJ. 2015 Feb 6;350:h391. doi: 10.1136/bmj.h391. No abstract available. PMID 25662947
- [Background] Copas AJ, Lewis JJ, Thompson JA, Davey C, Baio G, Hargreaves JR. Designing a stepped wedge trial: three main designs, carry-over effects and randomisation approaches. Trials. 2015 Aug 17;16:352. doi: 10.1186/s13063-015-0842-7. PMID 26279154
- [Background] Baio G, Copas A, Ambler G, Hargreaves J, Beard E, Omar RZ. Sample size calculation for a stepped wedge trial. Trials. 2015 Aug 17;16:354. doi: 10.1186/s13063-015-0840-9. PMID 26282553
- [Background] Hussey MA, Hughes JP. Design and analysis of stepped wedge cluster randomized trials. Contemp Clin Trials. 2007 Feb;28(2):182-91. doi: 10.1016/j.cct.2006.05.007. Epub 2006 Jul 7. PMID 16829207
- [Background] Hemming K, Taljaard M. Sample size calculations for stepped wedge and cluster randomised trials: a unified approach. J Clin Epidemiol. 2016 Jan;69:137-46. doi: 10.1016/j.jclinepi.2015.08.015. Epub 2015 Sep 5. PMID 26344808
- [Background] van den Ende C, Marano C, van Ahee A, Bunge EM, De Moerlooze L. The immunogenicity of GSK's recombinant hepatitis B vaccine in children: a systematic review of 30 years of experience. Expert Rev Vaccines. 2017 Aug;16(8):789-809. doi: 10.1080/14760584.2017.1338569. Epub 2017 Jul 3. PMID 28586278
- [Background] Jourdain G, Ngo-Giang-Huong N, Harrison L, Decker L, Khamduang W, Tierney C, Salvadori N, Cressey TR, Sirirungsi W, Achalapong J, Yuthavisuthi P, Kanjanavikai P, Na Ayudhaya OP, Siriwachirachai T, Prommas S, Sabsanong P, Limtrakul A, Varadisai S, Putiyanun C, Suriyachai P, Liampongsabuddhi P, Sangsawang S, Matanasarawut W, Buranabanjasatean S, Puernngooluerm P, Bowonwatanuwong C, Puthanakit T, Klinbuayaem V, Thongsawat S, Thanprasertsuk S, Siberry GK, Watts DH, Chakhtoura N, Murphy TV, Nelson NP, Chung RT, Pol S, Chotivanich N. Tenofovir versus Placebo to Prevent Perinatal Transmission of Hepatitis B. N Engl J Med. 2018 Mar 8;378(10):911-923. doi: 10.1056/NEJMoa1708131. PMID 29514030
- [Background] Collenberg E, Ouedraogo T, Ganame J, Fickenscher H, Kynast-Wolf G, Becher H, Kouyate B, Krausslich HG, Sangare L, Tebit DM. Seroprevalence of six different viruses among pregnant women and blood donors in rural and urban Burkina Faso: A comparative analysis. J Med Virol. 2006 May;78(5):683-92. doi: 10.1002/jmv.20593. PMID 16555290
- [Background] Hyams KC. Risks of chronicity following acute hepatitis B virus infection: a review. Clin Infect Dis. 1995 Apr;20(4):992-1000. doi: 10.1093/clinids/20.4.992. PMID 7795104
- [Background] Njai HF, Shimakawa Y, Sanneh B, Ferguson L, Ndow G, Mendy M, Sow A, Lo G, Toure-Kane C, Tanaka J, Taal M, D'alessandro U, Njie R, Thursz M, Lemoine M. Validation of rapid point-of-care (POC) tests for detection of hepatitis B surface antigen in field and laboratory settings in the Gambia, Western Africa. J Clin Microbiol. 2015 Apr;53(4):1156-63. doi: 10.1128/JCM.02980-14. Epub 2015 Jan 28. PMID 25631805
- [Background] Riou J, Ait Ahmed M, Blake A, Vozlinsky S, Brichler S, Eholie S, Boelle PY, Fontanet A; HCV epidemiology in Africa group. Hepatitis C virus seroprevalence in adults in Africa: a systematic review and meta-analysis. J Viral Hepat. 2016 Apr;23(4):244-55. doi: 10.1111/jvh.12481. Epub 2015 Oct 19. PMID 26477881
- [Background] Vray M, Debonne JM, Sire JM, Tran N, Chevalier B, Plantier JC, Fall F, Vernet G, Simon F, Mb PS. Molecular epidemiology of hepatitis B virus in Dakar, Senegal. J Med Virol. 2006 Mar;78(3):329-34. doi: 10.1002/jmv.20544. PMID 16419106
- [Background] Lemoine M, Shimakawa Y, Njie R, Taal M, Ndow G, Chemin I, Ghosh S, Njai HF, Jeng A, Sow A, Toure-Kane C, Mboup S, Suso P, Tamba S, Jatta A, Sarr L, Kambi A, Stanger W, Nayagam S, Howell J, Mpabanzi L, Nyan O, Corrah T, Whittle H, Taylor-Robinson SD, D'Alessandro U, Mendy M, Thursz MR; PROLIFICA investigators. Acceptability and feasibility of a screen-and-treat programme for hepatitis B virus infection in The Gambia: the Prevention of Liver Fibrosis and Cancer in Africa (PROLIFICA) study. Lancet Glob Health. 2016 Aug;4(8):e559-67. doi: 10.1016/S2214-109X(16)30130-9. PMID 27443781
- [Background] Duffy D, Mottez E, Ainsworth S, Buivan TP, Baudin A, Vray M, Reed B, Fontanet A, Rohel A, Petrov-Sanchez V, Abel L, Theodorou I, Miele G, Pol S, Albert ML. An in vitro diagnostic certified point of care single nucleotide test for IL28B polymorphisms. PLoS One. 2017 Sep 6;12(9):e0183084. doi: 10.1371/journal.pone.0183084. eCollection 2017. PMID 28877177
- [Background] Posuwan N, Payungporn S, Tangkijvanich P, Ogawa S, Murakami S, Iijima S, Matsuura K, Shinkai N, Watanabe T, Poovorawan Y, Tanaka Y. Genetic association of human leukocyte antigens with chronicity or resolution of hepatitis B infection in thai population. PLoS One. 2014 Jan 23;9(1):e86007. doi: 10.1371/journal.pone.0086007. eCollection 2014. PMID 24465836
- [Background] Demolis R, Botao C, Heyerdahl LW, Gessner BD, Cavailler P, Sinai C, Magaco A, Le Gargasson JB, Mengel M, Guillermet E. A rapid qualitative assessment of oral cholera vaccine anticipated acceptability in a context of resistance towards cholera intervention in Nampula, Mozambique. Vaccine. 2018 Oct 22;36(44):6497-6505. doi: 10.1016/j.vaccine.2017.10.087. Epub 2017 Nov 27. PMID 29174106
- [Background] Janzen J. The Social Fabric of Health: An Introduction to Medical Anthropology. McGraw-Hill; 2002.
- [Background] Winkelman M. Culture and Health: Applying Medical Anthropology. Jossey-Bass. 2008.
- [Background] Giles-Vernick T, Traore A, Bainilago L. Incertitude, Hepatitis B, and Infant Vaccination in West and Central Africa. Med Anthropol Q. 2016 Jun;30(2):203-21. doi: 10.1111/maq.12187. Epub 2016 Mar 31. PMID 25624042
- [Background] Scott S, Odutola A, Mackenzie G, Fulford T, Afolabi MO, Lowe Jallow Y, Jasseh M, Jeffries D, Dondeh BL, Howie SR, D'Alessandro U. Coverage and timing of children's vaccination: an evaluation of the expanded programme on immunisation in The Gambia. PLoS One. 2014 Sep 18;9(9):e107280. doi: 10.1371/journal.pone.0107280. eCollection 2014. PMID 25232830
- [Background] Briggs AH, Goeree R, Blackhouse G, O'Brien BJ. Probabilistic analysis of cost-effectiveness models: choosing between treatment strategies for gastroesophageal reflux disease. Med Decis Making. 2002 Jul-Aug;22(4):290-308. doi: 10.1177/0272989X0202200408. PMID 12150595
- [Derived] Tall H, Adam P, Tiendrebeogo ASE, Vincent JP, Schaeffer L, von Platen C, Fernandes-Pellerin S, Sawadogo F, Bokoum A, Bouda G, Ouattara S, Ouedraogo I, Herrant M, Boucheron P, Sawadogo A, Betsem E, Essoh A, Kabore L, Ouattara A, Meda N, Hien H, Gosset A, Giles-Vernick T, Boyer S, Kania D, Vray M, Shimakawa Y. Impact of Introducing Hepatitis B Birth Dose Vaccines into the Infant Immunization Program in Burkina Faso: Study Protocol for a Stepped Wedge Cluster Randomized Trial (NeoVac Study). Vaccines (Basel). 2021 Jun 1;9(6):583. doi: 10.3390/vaccines9060583. PMID 34206058